CLINICAL TRIAL: NCT01227252
Title: Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY2886721 in Healthy Subjects
Brief Title: A Safety Study of LY2886721 Multiple Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13734; I4O-MC-BACB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2886721 (Experimental)
  Interventions: Drug: LY2886721
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2886721 — 5 milligrams (mg) up to 35 mg, administered orally as capsules, daily for 14 days
  Arms: LY2886721
Drug: Placebo — Administered orally as capsules, daily for 14 days
  Arms: Placebo

SUMMARY:
This is a Phase 1 study in healthy subjects to evaluate the safety and tolerability of LY2886721 multiple doses, how the body handles the drug, and the drug's effect on the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-childbearing potential women
* Body mass index between 18.0-32.0 kilograms per square meter (kg/m^2)
* Are reliable and willing to make yourself available for the duration of the study and are willing to follow study procedures and research unit policies

Exclusion Criteria:

* Taking over-the-counter or prescription medication with the exception of vitamins or minerals
* Smoke more than 10 cigarettes per day
* Drink more than 5 cups of caffeine containing beverages (for example, coffee, tea) per day

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo was administered orally as capsules, once daily for 14 days.
- 5 mg LY2886721: A 5-milligram (mg) dose of LY2886721 was administered orally as capsules, once daily for 14 days.
- 15 mg LY2886721: A 15-mg dose of LY2886721 was administered orally as capsules, once daily for 14 days.
- 35 mg LY2886721: A 35-mg dose of LY2886721 was administered orally as capsules, once daily for 14 days.
Period: Overall Study
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Started | 12 | 10 | 10 | 10
Received at Least 1 Dose of Study Drug | 12 | 10 | 10 | 10
Completed | 12 | 7 | 10 | 10
Not Completed | 0 | 3 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721 | Total
Number analyzed (Participants) | 12 | 10 | 10 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 10 | 10 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 3
  Male | 12 | 9 | 9 | 9 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 2 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 1 | 8
  White | 6 | 3 | 5 | 6 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 10 | 10 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and nonserious adverse events. A summary of serious and all other nonserious adverse events is located in the Reported Adverse Event module. The number of participants with at least 1 adverse event in each treatment arm is reported for this outcome measure.
Time Frame: Predose up to Day 70
Population: All randomized participants were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 12 | 10 | 10 | 10
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0
  Nonserious Adverse Events | 2 | 2 | 3 | 3

2. Secondary Outcome: Plasma Maximum Observed Drug Concentration at Steady State (Cmax,ss) of LY2886721
Time Frame: Predose (Day 14) up to Day 19
Population: All participants who received study drug on Day 14 and had evaluable pharmacokinetic data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 5 mg LY2886721: Participants received a 5-mg oral dose of LY2886721 capsules, once daily for 14 days.
- 15 mg LY2886721: Participants received a 10-mg oral dose of LY2886721 capsules, once daily for 14 days.
- 35 mg LY2886721: Participants received a 35-mg oral dose of LY2886721 capsules, once daily for 14 days.
Arm/Group | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 9 | 10 | 10
nanogram per milliliter (ng/mL) | 11.6 (48) | 43.0 (24) | 80.0 (43)

3. Secondary Outcome: Plasma Area Under the Concentration Versus Time Curve (AUC) of LY2886721
Description: Area under the concentration versus time curve during 1 dosing interval (1 dosing interval=24 hours) at steady state (AUCτ,ss) is being reported for this outcome measure.
Time Frame: Predose (Day 14) to 24 Hours post-dose (Day 15)
Population: All participants who received study drug on Day 14 and had evaluable pharmacokinetic data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 9 | 10 | 10
nanogram*hour per milliliter (ng*h/mL) | 128 (41) | 447 (23) | 861 (38)

4. Secondary Outcome: Plasma Amyloid Beta (Aβ) 1-40 Concentration
Description: The minimum concentration (Cnadir) is being reported for this outcome measure.
Time Frame: Predose (Day 14) up to Day 19
Population: All participants who received study drug on Day 14 and had evaluable pharmacodynamic data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 12 | 9 | 10 | 10
picogram per milliliter (pg/mL) | 123 (14.5) | 49 (55.1) | 40 (19.7) | 25 (28.1)

5. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentration of LY2886721
Time Frame: 24 Hours post-dose (Day 15)
Population: A subset of all participants who received study drug on Day 14 and had evaluable pharmacodynamic data was included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 4 | 4 | 4
nanogram per milliliter (ng/mL) | 0.5 (64.5) | 1.4 (16.6) | 3.8 (22.6)

6. Secondary Outcome: Change From Baseline to Day 15 Endpoint in Cerebrospinal Fluid (CSF) Amyloid Beta (Aβ) 1-40 Concentration
Description: The Least Squares means were adjusted for baseline concentration.
Time Frame: Predose (Day 14), 24 Hours post-dose (Day 15)
Population: All participants who received study drug on Day 14 and had evaluable pharmacodynamic data were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change (%)
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Number analyzed (Participants) | 12 | 10 | 10 | 10
percent change (%) | -3.9 [-9.1 to 1.3] | -11.8 [-16.1 to -7.4] | -27.5 [-31.6 to -23.5] | -59.1 [-67.0 to -51.1]

ADVERSE EVENTS:
Arm/Group | Placebo | 5 mg LY2886721 | 15 mg LY2886721 | 35 mg LY2886721
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/12 | 2/10 | 3/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | 5 mg LY2886721 (N=10) | 15 mg LY2886721 (N=10) | 35 mg LY2886721 (N=10)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual field tests abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days